CLINICAL TRIAL: NCT07357675
Title: A Clinical Trial To Investigate The Effect Of EA-230 On Hospital Length of Stay In Patients With Coronary Artery Disease (CAD) Undergoing Coronary Artery Bypass Grafting (CABG) Surgery.
Acronym: EasyBoost
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EBI Anti Sepsis BV (Industry)
Collaborators: CR2O B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EasyBoost
Record Dates: First submitted 2026-01-16; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease (CAD); Coronary Artery Bypass Graft Surgery(CABG)
MeSH Terms: conditions — Coronary Artery Disease | interventions — alanyl-glutaminyl-glycyl-valine

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Phase III Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EA-230 90mg/kg/hour (Experimental)
  Interventions: Drug: EA-230 90mg/kg/hour
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EA-230 90mg/kg/hour — Intravenous administration of 90mg/kg per hour for 4 hours.
  Arms: EA-230 90mg/kg/hour
Drug: Placebo — Placebo administered intravenously for 4 hours
  Arms: Placebo

SUMMARY:
EA-230 is a new therapy that may help people recover faster and have fewer problems after bypass surgery. In an earlier clinical trial, participants who received EA-230 during Coronary Artery Bypass surgery stayed in the Intensive Care Unit (ICU) and the hospital for a shorter time and had fewer serious complications, compared to those who received a placebo (an inactive therapy). The use of EA-230 was safe and well tolerated. This trial will test EA-230 in more participants to see if it really works and is safe to use in the future.

This is a Phase III trial. It will take place in multiple locations and will follow a double-blind, randomized, placebo-controlled clinical design, meaning neither doctors nor participants will know whether they receive EA-230 or placebo during the trial. Assignment to EA-230 or placebo occurs by chance, like throwing dice. The total duration of the trial, including medical check-ups, will be approximately 71 days. There is a total of 10 visits, including a screening-, a pre-operative-, and 2 remote visits. 7 of these visits are during your stay at the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years, both male and female.
2. Patients scheduled for elective on-pump CABG with at least 3 bypasses, with or without valve replacement.
3. For women of childbearing potential (WOCBP), agree to use adequate contraception17 from enrollment and up to 28 days after IMP administration, and must have a negative pregnancy test prior to entry into the trial.
4. For male patients, agree to use adequate contraception and refrain from donating sperm from enrollment and up to 28 days after IMP administration.
5. Willing and able to give written informed consent.

Exclusion Criteria:

1. Patients undergoing non-elective on-pump CABG (i.e., emergency surgery). Emergency surgery is defined as planned surgery within 24 hours of diagnosis.
2. Cardiogenic shock or hemodynamic instability that requires inotropes, vasopressors, or other mechanical devices, such as an intra-aortic balloon counter-pulsation (IABP), within 24 hours prior to surgery.
3. Use of a left ventricular assist device (LVAD), or intra-aortic balloon pump or other cardiac devices, within 7 days prior to surgery.
4. A requirement for any of the following within 7 days prior to surgery: defibrillator or permanent pacemaker, mechanical ventilation, IABP, LVAD, or other forms of mechanical circulatory support.
5. Required cardiopulmonary resuscitation within 14 days prior to cardiac surgery.
6. Known chronic liver disorder with Child-Pugh C classification.
7. Confirmed or treated endocarditis requiring antimicrobial or antiviral treatment within 30 days prior to surgery or other current active infection requiring antimicrobial or antiviral treatment within 14 days prior to surgery.
8. Ongoing sepsis (as defined by SEPSIS-3) within 2 weeks of screening or, in the opinion of the investigator, an untreated clinically significant infection (viral or bacterial) prior to or at Screening and before randomization.
9. Immuno-compromised patients, as self-reported or as observed in medical records, including patients:

   1. with solid organ transplantation.
   2. known to be positive for human immunodeficiency virus (HIV).
   3. that use immunosuppressive drugs or have received recent chemotherapy, at the discretion of the Investigator and including patients;

   i. with active malignancy who have undergone chemotherapy within 30 days prior to trial entry.

   ii. receiving chronic corticosteroid treatment equivalent to a prednisone dose of 10 mg or higher per day, within 30 days prior to trial entry, or an equivalent dose of another corticosteroid or any other anti-inflammatory or inflammation-suppressing medications such as interleukin blockers, methotrexate or similar therapies. Non-Steroidal Anti-Inflammatory Drugs are not exclusionary.
10. Patients with hematological disorders (known disorders from myeloid and/or lymphoid origin, leucopenia (both active and in remission)).
11. Known severe renal disease requiring dialysis, or a known estimated Glomerular Filtration Rate (eGFR) prior to admission of < 20 ml/min/1.73 m2.
12. Women who are pregnant, breastfeeding or planning to become pregnant during the trial or within 28 days after IMP administration.
13. Previous receipt of EA-230.
14. Known hypersensitivity to the IMP.
15. Use of any investigational drug within 1 month or 5 half-lives of said investigational drug (whichever is longer) prior to IMP administration in this trial. Participation in an observational clinical trial is not exclusionary.
16. Patients (or partners of patients) not willing to use a reliable method of contraception from enrollment and up to 28 days after IMP administration.
17. Patients who are unable to communicate effectively in the local language of the trial site, at the discretion of the Investigator.
18. Inability to personally provide written informed consent.
19. Known or suspected of not being able to comply with the trial protocol, at the discretion of the Investigator.
20. Any other condition which, in the Investigator's opinion, will interfere with completion of the trial.
21. Being an employee of the Investigator or trial site with direct involvement in the proposed trial or other studies under the direction of that Investigator or trial site or being a family member of an employee of the Investigator with direct involvement in the proposed trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-03-24 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Required postoperative hospital length of stay | Up to 28 days
  Median postoperative duration, from the moment of first incision until the time when a patient is eligible to be discharged from the hospital.

SECONDARY OUTCOMES:
Required postoperative ICU length of stay | Up to 28 days
  Median postoperative duration, from the moment of first incision until the time when a patient is eligible to be discharged from the ICU and transferred to the general ward.
Actual postoperative hospital length of stay | Up to 28 days
  Median postoperative duration, from the moment of first incision until the time when a patient is actually discharged from the hospital.
Actual postoperative ICU length of stay | Up to 28 days
  Median postoperative duration, from the moment of first incision until the time when a patient is actually discharged from the ICU and transferred to the general ward.
Single Organ Outcome Measures (SOOMs) | Up to 28 days
  Median cumulative duration of moderate and severe Single Organ Outcome Measures (SOOMs) according to the European Perioperative Clinical Outcome (EPCO) definitions during the trial.
Net Fluid Balance (NFB) in milliliters (mL) | Up to 2 days (48 hours) after start of surgery (first incision)
  Median cumulative NFB at the start of IMP administration (T0) and up to 24 and 48 hours thereafter. NFB is measured by the difference between a patient's total fluid intake and total fluid output. This includes all intravenous fluids, oral intake, and nutritional feeds against urine output, drainage, and other fluid losses. No correction is applied for insensible losses (e.g., sweating, or respiratory exhalation).
Vasopressor use in microgram per kilogram (µg/kg) and/or international units (IU) | Up to 2 days (48 hours) after start of surgery (first incision)
  Cumulative dose of vasopressors at the start of IMP administration (T0) and up to 24 and 48 hours thereafter.
Inotropic use in microgram per kilogram (µg/kg) | Up to 2 days (48 hours) after start of surgery (first incision)
  Cumulative dose of inotropes at the start of IMP administration (T0) and up to 24 and 48 hours thereafter.
Vasopressor-Inotropic Score | Up to 2 days (48 hours) after start of surgery (first incision)
  Vasopressor-inotropic score at the start of IMP administration (T0) and up to 24 and 48 hours thereafter.
  Vasoactive-Inotropic Score is calculated as follows: Dopamine dose (µg/kg/min) + Dobutamine dose (µg/kg/min) + 100 * Epinephrine dose (µg/kg/min) + 100 * Norepinephrine dose (µg/kg/min) + 100 * Vasopressin dose (units/min) + 1000 * Milrinone dose (µg/kg/min) + 2000 * Levosimendan dose (µg/kg/min).
Blood plasma levels of EA-230 in microgram per liter (µg/L) | Up to 4 hours after IMP administration (on Day 1)
  Blood plasma levels of EA-230 measured immediately before the end of EA-230 infusion (T4) in all patients.
  Blood plasma levels of EA-230 measured at T0, T0.5, T1, T2, T3 and T4 in a subset of patients in the Netherlands.
  Only venous blood is sampled to determine blood plasma levels.
Treatment emergent (Serious) Adverse Events and Adverse Drug Reactions | Up to 28 days
  Incidence of treatment emergent (Serious) Adverse Events and Adverse Drug Reactions during the trial period. Coded using the Medical Dictionary for Regulatory Activities (version 28 or higher) and graded according to the Common Terminology Criteria for Adverse Events (V6.0).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickers, Prof., Principal Investigator — Radboudmc
Locations (5):
- MAYO clinic, Rochester, Minnesota, United States
- UZ Gent, Ghent, Belgium
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede
  - RadboudUMC, Nijmegen
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The IPD might be shared in the future, this is currently undecided. This field will be updated in case the data will be shared in the future.